CLINICAL TRIAL: NCT05375747
Title: Comparison Between Remimazolam Versus Propopol Based Total Intravenous Anesthesia for Breast Surgery : a Randomized Controlled Trial
Brief Title: Remimazolam Versus Propopol Based Total Intravenous Anesthesia for Breast Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants due to hospital conditions
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seokha Yoo, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2112-150-1286
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam based total intravenous anesthesia (Experimental): For induction and maintenance of anesthesia, total intravenous anesthesia is performed using continuous intravenous infusion of remimazolam and remifentanil.
  Interventions: Drug: Remimazolam
- Propofol based total intravenous anesthesia (Active Comparator): For induction and maintenance of anesthesia, total intravenous anesthesia is performed using continuous intravenous infusion of propofol and remifentanil.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — For induction and maintenance of anesthesia, total intravenous anesthesia is performed using continuous intravenous infusion of remimazolam and remifentanil.
  Arms: Remimazolam based total intravenous anesthesia
Drug: Propofol — For induction and maintenance of anesthesia, total intravenous anesthesia is performed using continuous intravenous infusion of propofol and remifentanil.
  Arms: Propofol based total intravenous anesthesia

SUMMARY:
Comparison of the incidence of hypotension under remimazolam and propofol-based anesthesia in patients undergoing breast surgery under general anesthesia

DETAILED DESCRIPTION:
The purpose of this study was to investigate whether remimazolam-based general anesthesia could reduce the incidence of hypotension in patients undergoing breast surgery under general anesthesia compared to propofol-based general anesthesia. The purpose of this study is to establish and test the hypothesis that the incidence of hypotension under general anesthesia based on remimazolam will be less than that of propofol based general anesthesia. In addition, this study compares the proportion of patients who require a vasopressor, the time taken for anesthesia induction, the time to recover from anesthesia, postoperative pain, the incidence of postoperative nausea and vomiting, the quality of postoperative recovery, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 19 undergoing elective breast cancer surgery under general anesthesia at Seoul National University Hospital

Exclusion Criteria:

* patients with acute narrow-angle glaucoma/ shock or coma/ acute alcohol poisoning/ sleep apnea/ alcohol or drug dependency/ severe or acute respiratory failure/ galactose intolerance/ Lapp lactase deficiency/ glucose galactose malabsorption/ severe hypersensitivity to dextran.
* Patients with myasthenia gravis/ pulmonary heart disease/ chronic obstructive pulmonary disease/ bronchial asthma
* Patients with cardiovascular diseases such as ischemic heart disease/ coronary artery disease/ angina pectoris/ myocardial infarction/ atherosclerosis/ arrhythmia/ cerebrovascular disease/ and stroke
* Patients with chronic renal failure
* Patients with severe hepatic impairment (Child Pugh class C)
* Patients with American Society of Anesthesiology score III or higher
* Patients with hypersensitivity to propofol and soy or peanuts
* Epilepsy patients
* Patient with fat metabolism abnormality
* Patients with high intracranial pressure
* Pregnant woman
* Patients unable to use supraglottic airway due to poor dental condition
* In cases that the researcher judges to be unsuitable for this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Hypotension incidence | from induction of anesthesia to end of surgery
  Incidence of hypotension (MAP <65 mmHg) from induction of anesthesia to end of surgery

SECONDARY OUTCOMES:
Use of vasopressor | from induction of anesthesia to end of surgery
  Proportion of patients using vasopressors due to hypotension from induction of anesthesia to completion of surgery
Number of occurrences of hypotension during surgery | from induction of anesthesia to end of surgery
  Number of occurrences of hypotension during surgery
Type of vasopressor used | from induction of anesthesia to end of surgery
  Type of vasopressor used
Total dose of vasopressor used | from induction of anesthesia to end of surgery
  Total dose of vasopressor used
Blood pressure | from induction of anesthesia to end of surgery
  Blood pressure during operation, noninvasive blood pressure is measured at lower leg
Heart rate | from induction of anesthesia to end of surgery
  Heart rate during operation
Saturation of percutaneous oxygen (SpO2) | from induction of anesthesia to end of surgery
  Saturation of percutaneous oxygen (SpO2) during operation
Patient State Index (PSi) | from induction of anesthesia to end of surgery
  Patient State Index (PSi) during operation
Incidence of bradycardia | from induction of anesthesia to end of surgery
  Incidence of bradycardia during operation, bradycardia is defined as heart rate less than 50
Severity of injection pain | At the start of induction of general anesthesia
  Severity of injection pain of sedative(propofol or remimazolam depending on group assignment) during induction of anethesia: none/ mild/ moderate/ severe
Incidence of intraoperative awareness | from induction of anesthesia to end of surgery
  Incedence of intraoperative awareness during operation
Incidence of intraoperative body movement | from induction of anesthesia to end of surgery
  Incidence of intraoperative body movement during operation
Incidence of use of rescue sedative agents | from induction of anesthesia to end of surgery
  Incidence of use of any kinds of rescue sedative agents
T ime from start of administration of sedative drug to loss of consciousness | from induction of anesthesia to loss of consciousness
  T ime from start of administration of sedative drug to loss of consciousness
Time from the end of administration of sedative to eye opening | from end of administration of sedative to eye opening
  Time from the end of administration of sedative(propofol or remimazolam depending on group assignment) to eye opening
Time from the end of administration of sedative to response to verbal command | from end of administration of sedative to response to verbal command
  Time from the end of administration of sedative(propofol or remimazolam depending on group assignment) to response to verbal command
Time from the end of administration of sedative to supraglottic airway removal | from end of administration of sedative to supraglottic airway removal
  Time from the end of administration of sedative(propofol or remimazolam depending on group assignment) to supraglottic airway removal
Duration of post anesthesia care unit stay | From entering post anesthesia care unit until leaving, post-operatively 1 hour average
  Duration of post anesthesia care unit stay
Total analgesic consumption for 24 hours after surgery | For 24 hours after the end of surgery
  Total analgesic consumption for 24 hours after surgery
Numeric rating scale score in the recovery room immediately after surgery | Immediate after end of surgery
  Numeric rating scale score in the recovery room immediately after surgery, Numeric rating scale: 0 points for no pain, 10 points for the worst pain imaginable / The higher the number, the more severe the pain
Incidence of nausea and vomiting within 24 hours after surgery | within 24 hours after surgery
  Incidence of nausea and vomiting within 24 hours after surgery
Severity of nausea and vomiting within 24 hours after surgery | within 24 hours after surgery
  Severity of nausea and vomiting within 24 hours after surgery: none,. mild, moderate, severe
Subjective sleep quality on the day of surgery | During the day of surgery
  Subjective sleep quality on the day of surgery, Score out of 10, the higher the number, the better the quality of sleep
Patient satisfaction with anesthesia | The day of operation
  Patient satisfaction with anesthesia, Score out of 10, the higher the number, the better the quality of sleep
Hospital length of stay | From administration to discharge, average 4 days
  Hospital length of stay
15 item Quality of Recovery | 24 hours after surgery
  15 item Quality of Recovery: 15-item questionnaire about the degree of recovery after surgery, 10 points per question, total 150 points

CONTACTS AND LOCATIONS:
Overall Officials: Seokha Yoo, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No